CLINICAL TRIAL: NCT03197389
Title: Effect of Pembrolizumab (Keytruda®) on Biomarkers Related to Intratumoral Immunity, Proliferation and Apoptosis in Early Breast Cancer.
Brief Title: Effect of Pembrolizumab (Keytruda®) on Biomarkers in Early Breast Cancer.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MK 3475-318
Record Dates: First submitted 2017-06-02; First posted 2017-06-23 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Hormone Receptor Negative Neoplasm
Keywords: Biomarker
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort A1 (Other): Cohort A1 will include patients with a triple negative breast tumor. Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab
- Cohort A2 (Other): Cohort A2 will include patients with ER/PR negative and Her2 positive breast tumor. Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab
- Cohort B1 (Other): Cohort B1 will include patients with a triple negative breast tumor who received neoadjuvant chemotherapy and who have clear signs of residual tumor on imaging after finishing neoadjuvant chemotherapy (i.e. on imaging estimated residual tumor size of at least 10 mm). Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab
- Cohort B2 (Other): Cohort B2 will include patients with a ER/PR negative and Her2 positive breast tumor who received neoadjuvant chemotherapy and who have clear signs of residual tumor on imaging after finishing neoadjuvant chemotherapy (i.e. on imaging estimated residual tumor size of at least 10 mm). Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab
- Cohort A3 (Other): Cohort A3 will include patients with ER positive breast tumor. Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab
- Cohort B3 (Other): Cohort B3 will include patients with a ER positive breast tumor who received neoadjuvant chemotherapy and who have clear signs of residual tumor on imaging after finishing neoadjuvant chemotherapy (i.e. on imaging estimated residual tumor size of at least 10 mm). Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Biological: humanized anti-PD-1 monoclonal antibody humanized anti-PD-1 monoclonal antibody is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda

SUMMARY:
The study consists of 2 parts: a retrospective study, and a prospective clinical study with pembrolizumab (Keytruda®) (Phase 0).

1. Retrospective study (S58910):

   This is a retrospective analysis to study the expression of PD-L1 in ER/PR negative breast tumors and to correlate this PD-L1 expression with tumor infiltrating lymphocytes (TILs), proliferation, expression of apoptosis and clinical outcome (development of distant metastases).
2. Phase 0 study:

This is a Phase 0 single center, open-label, non-randomized, study in patients with early breast cancer. Patients will be treated with one injection of Pembrolizumab (Keytruda®) administered intravenously at 200 mg 10 +/- 4 days before surgery. This phase 0 study will consist of 2 cohorts; cohort A will include patients who are scheduled for upfront surgery. Cohort A1 will include patients with Her2 negative tumors, Cohort A2 patients with Her2 positive tumors and Cohort A3 with ER positive tumours. Cohort B will include patients who received neoadjuvant chemotherapy (with anti-Her2 therapy if Her2 positive) and who have clear signs of residual tumor on imaging after finishing neoadjuvant chemotherapy (i.e. on imaging estimated residual tumor size of at least 10 mm). Cohort B1 will include Her2 negative tumors, Cohort B2 Her2 positive tumors and Cohort B3 ER positive tumors. The injection will be given in the oncological outpatient unit. Patients will be monitored carefully for the development of adverse experiences/events. Adverse experiences/events will be evaluated according to criteria outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion if needed. Newly obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 0. Subjects for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
4. Have a performance status of 0 or 1 on the ECOG Performance Scale.
5. Have non-metastatic operable newly diagnosed primary invasive carcinoma of the breast that is:

   1. Histologically confirmed
   2. ER/PR negative or ER positive. ER/PR status will be evaluated with Allred score (semi-quantitative measurement) following ASCO CAP guidelines 2009.
   3. HER2 negative of positive. HER2 status will be evaluated using IHC followed by FISH with dual probe (ASCO CAP guidelines 2013).
   4. Primary tumor size greater than 1 cm, measured by any of clinical examination, mammography, ultrasound or magnetic resonance imaging
   5. Any clinical nodal status
6. Have evaluable core biopsy for IHC
7. Be willing to provide plasma/blood samples
8. After neo-adjuvant chemotherapy (cohort B1 and B2) patients must have residual tumor >1cm and must be willing to provide evaluable new tumor biopsy for IHC
9. Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after receiving the study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, until 120 after receiving the study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of receiving the treatment dose.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to receiving the trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 0 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent or co-inhibitory T-cell receptor therapy (e.g. OX40-CD137, CTLA-4)
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Smeets, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort B1 | Cohort B2 | Cohort B3
Started | 16 | 5 | 18 | 9 | 1 | 5
Completed | 16 | 5 | 18 | 9 | 1 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort B1 | Cohort B2 | Cohort B3 | Total
Number analyzed (Participants) | 16 | 5 | 18 | 9 | 1 | 5 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 15 | 7 | 1 | 3 | 40
  >=65 years | 6 | 1 | 3 | 2 | 0 | 2 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 18 | 9 | 1 | 5 | 54
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 16 | 5 | 18 | 9 | 1 | 5 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 16 | 5 | 18 | 9 | 1 | 5 | 54

OUTCOME MEASURES:

1. Primary Outcome: PD-1 Expression
Description: PD-1 expression after a single dose of pembrolizumab.
  Immunohistochemical stains were performed on 5-μm thick sections using an automatic immunostainer (Bond Max Autostainer, Leica) according to the manufacturer's instructions.
  A monoclonal antibodie was used for PD1 (clone NAT105, Abcam). PD1 expression on sTIL was assessed semi quantitatively.
Time Frame: 2 years
Population: The overall number of participants analyzed is not consistent with the numbers provided in any of the rows in the participant flow module because it was not always possible to interpret all the immunohistochemical stainings of all patients due to bad quality of the study samples.
Measure: Median (Full Range); unit: percentage
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort B1 | Cohort B2 | Cohort B3
Number analyzed (Participants) | 15 | 4 | 14 | 6 | 1 | 3
percentage | 0 [0 to 10] | 0 [0 to 1] | 0 [0 to 5] | 0 [0 to 5] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Cohort A1 vs Cohort A2 vs Cohort A3 vs Cohort B1 vs Cohort B2 vs Cohort B3; Test type: Other; Median Difference (Net) = 0

ADVERSE EVENTS:
Time Frame: Adverse events were actively reviewed at 10 +/- 4 days and 30 +/- 7 days after administration of the study medication.
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort B1 | Cohort B2 | Cohort B3
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/5 | 0/18 | 0/9 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/5 | 0/18 | 0/9 | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/16 | 0/5 | 0/18 | 0/9 | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03197389/Prot_SAP_000.pdf